CLINICAL TRIAL: NCT02878421
Title: Vascular Effects of Regular Cigarettes Versus electronIc Cigarette Use
Acronym: VESUVIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); British Heart Foundation (Other)
Responsible Party: Principal Investigator, Professor. Jacob George, Professor, University of Dundee
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2014CV10
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Vascular Diseases
MeSH Terms: conditions — Vascular Diseases | interventions — Tobacco Use Cessation Devices; Electronic Nicotine Delivery Systems; Nicotine; Flavoring Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- tobacco cigarette (Active Comparator): Intervention: tobacco cigarettes min 15/day
  Interventions: Other: Tobacco cigarette
- e.cigarettes + 16mg nicotine & flavor (Active Comparator): Intervention: One flavoured electronic cigarette 16mg nicotine/day
  Interventions: Device: electronic cigarette + 16mg nicotine & flavor
- e.cigarettes + 0mg nicotine & flavour (Active Comparator): Intervention: One electronic cigarette with flavour +0mg nicotine/day
  Interventions: Other: electronic cigarette + 0mg nicotine & flavor

INTERVENTIONS:
Device: electronic cigarette + 16mg nicotine & flavor — comparison of different strengths of nicotine
  Other Names: vapourlites; e.cigarette
  Arms: e.cigarettes + 16mg nicotine & flavor
Other: electronic cigarette + 0mg nicotine & flavor — comparison of different strengths of nicotine
  Other Names: vapourlites; e.cigarette
  Arms: e.cigarettes + 0mg nicotine & flavour
Other: Tobacco cigarette — Participant to remain on traditional cigarettes for 28 days
  Other Names: Traditional cigarette, any brand
  Arms: tobacco cigarette

SUMMARY:
The purpose of this study is to assess the effects of electronic cigarettes-nicotine and electronic cigarette-nicotine free on endothelial function as compared to traditional cigarettes. Due to ethical reasons, we cannot fully randomise all particpants to the three arms.

Participants who wish to quit smoking will be randomized to

1. Switch to electronic cigarettes containing nicotine plus flavor
2. Switch to electronic cigarettes containing flavor alone Those who do not wish to quit smoking will continue on the Tobacco Cigarette arm Treatment period will be 28 days

DETAILED DESCRIPTION:
Electronic cigarettes (EC) are gaining popularity as an alternative to Traditional Cigarettes (TC). Despite not containing all the harmful substances seen in TC, EC are known to contain impurities that may have a detrimental impact on human health. The effects of ECs compared with TC on vascular function, inflammation and oxidative stress are unknown. It is increasingly recognised that nicotine itself has significant atherothrombotic effects. Therefore, clinicians are unable to confidently recommend ECs as a less risky alternative to TC.

Hypothesis: Endothelial function will be improved on EC compared to TC when measured by flow mediated dilatation (FMD).

Potential benefit: This study will provide further information on the potential use these devices and the risks and/or benefits associated with them, specifically in relation to vascular health.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and over
* Currently smoking ≥15 full strength tobacco cigarettes per day for at least 2 years, or roll-up tobacco equivalent (cigar or pipe smokers not included).
* Willing to stop tobacco cigarettes for period of study if required
* Willing not to use electronic cigarettes if required
* Able to give informed consent

Exclusion Criteria:

* Pregnant or lactating.
* Women of childbearing potential who do not abstain from sex or use effective contraception.
* On current prescribed medication for cardiovascular disease.
* History of cardiovascular disease (excluding hypertension), diabetes, active malignance or chronic renal disease.
* Nut allergy
* Participation in another clinical trial (other than observational trials and registries) with an investigational product and/or intervention within 30 days before visit 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-08-18 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Flow mediated Dilation (FMD) between the TC group and the EC-nicotine and EC-nicotine free groups | Baseline and 1 month

SECONDARY OUTCOMES:
Change in FMD between EC-nicotine and EC-nicotine free groups | Baseline and 1 month
Change in FMD between TC and EC groups combined | Baseline and 1 month
Change in oxidised LDL between the TC, EC-nicotine free and EC-nicotine groups | Baseline and 1 month
Change in PAI-1 between the TC, EC-nicotine free and EC-nicotine groups | Baseline and 1 month
Change in hs-CRP between the TC, EC-nicotine free and EC-nicotine groups | Baseline and 1 month
Change in Pulse Wave Velocity between the TC group and the EC-nicotine free groups. | Baseline and 1 month
Change in tPA between the TC, EC-nicotine free and EC-nicotine groups | Baseline and 1 month
Change in Augmentation Index@75bpm between the TC group,EC-nicotine and the EC-nicotine free groups | Baseline and 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Jacob George, Principal Investigator — University of Dundee
Locations (1):
- University of Dundee, Dundee, Tayside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] George J, Hussain M, Vadiveloo T, Ireland S, Hopkinson P, Struthers AD, Donnan PT, Khan F, Lang CC. Cardiovascular Effects of Switching From Tobacco Cigarettes to Electronic Cigarettes. J Am Coll Cardiol. 2019 Dec 24;74(25):3112-3120. doi: 10.1016/j.jacc.2019.09.067. Epub 2019 Nov 15. PMID 31740017

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02878421/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT02878421/SAP_001.pdf